CLINICAL TRIAL: NCT02545972
Title: A Prospective Non-randomized Trial of Conversion From Twice a Day Tacrolimus to Once Daily Modified Release Tacrolimus
Brief Title: Once-a-day Tacrolimus Conversion Study: The OneTAC Trial
Acronym: OneTAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newark Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, David A. Baran, MD, Director, Heart Failure & Transplant Research, Newark Beth Israel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OneTAC
Record Dates: First submitted 2015-09-07; First posted 2015-09-10 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Heart Failure
Keywords: immunosuppression
MeSH Terms: conditions — Heart Failure | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Once a day tacrolimus (Experimental): Tacrolimus extended release will be given at an initial once daily dose equivalent to the total daily dose of the twice a day Tacrolimus formulation.
  Interventions: Drug: tacrolimus extended release

INTERVENTIONS:
Drug: tacrolimus extended release — daily dosing of tacrolimus
  Other Names: Astagraf

SUMMARY:
This study investigates the use of tacrolimus extended release in stable patients who have undergone a heart transplant. All patients will receive the study medication free of charge for the 1 year duration of the study.

DETAILED DESCRIPTION:
Tacrolimus has been extensively studied in solid organ transplantation. It is FDA approved for heart transplant recipients as a twice a day formulation (Prograf brand name, as well as generic formulations). A modified release formulation is available and FDA approved for kidney transplant recipients (Astagraf, Astellas Pharmaceutical), but is not approved for heart transplant patients.

In this study the investigators will study 100 patients who are stable on twice a day Tacrolimus and convert these subjects to once a day modified release Tacrolimus. The investigators will observe these patients for 1 year following the switch and assess safety and efficacy in a heart transplant population.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 or higher
* Heart transplant recipient at least 365 days post-transplant at time of study screening
* Informed consent available
* Willingness to return for study visits, clinically indicated bloodwork
* On tacrolimus-based chronic immunosuppression.
* Self-identified ethnic group is provided

Exclusion Criteria:

* Prior heart or solid organ transplant
* Less than 365 days post-transplant at study screening
* Receiving cyclosporine based immunosuppression or calcineurin inhibitor free regimen
* Concurrent kidney or other solid organ
* Inability to provide informed consent
* More than 15 years post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The change in glomerular filtration rate slope between the 6 months prior to study enrollment and 6 months post-study enrollment. | 6 months
  The change in the slope of the Glomerular filtration rate at 6 months prior to study enrollment as compared to 6 months post study enrollment

SECONDARY OUTCOMES:
The change in glomerular filtration rate slope between the 6 months prior to study enrollment and 12 months post-study enrollment. | 12 months
  The change in the slope of the Glomerular filtration rate at 6 months prior to study enrollment as compared to 12 months post study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David A Baran, MD, Principal Investigator — Newark Beth Israel Medical Center
Locations (1):
- Newark Beth Israel Medical Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No